CLINICAL TRIAL: NCT06366074
Title: Early-feasibility Study to Evaluate Usability and Safety of the Watch-Transcutaneous Electrical Acustimulation (TEA) Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not funded.
Sponsor: University of Michigan (Other)
Collaborators: Transtimulation Research, Inc (Other)
Responsible Party: Principal Investigator, Jiande Chen, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HUM00252120
Record Dates: First submitted 2024-04-01; First posted 2024-04-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Usability; Early feasibility; Safety

STUDY DESIGN:
Intervention Model Description: Prevalence of delayed Chemotherapy-induced nausea, emesis, and dyspeptic symptoms (CINEDS) is 75% in women vs 51% in men (60% to 40% ratio). Therefore, every effort will be made to recruit at least 60% female subjects into the clinical study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Watch-TEA (Experimental)
  Interventions: Device: Watch-TEA group; Device: Tethered TEA device
- Tethered TEA device (Experimental)
  Interventions: Device: Watch-TEA group; Device: Tethered TEA device

INTERVENTIONS:
Device: Watch-TEA group — Subjects will wear the device for 3 days. The subjects will self-apply the TEA for 60 min once daily with the current amplitude set at a maximal tolerable level.
  To increase the subject compliance, two measures will be implemented: timely alerts by the app (and phone calls, if needed) for performing the TEA sessions, and recording full history of therapy sessions on the device for monitoring the compliance.
Device: Tethered TEA device — Subjects will wear the device for 3 days. The subjects will self-apply the TEA for 60 min once daily with the current amplitude set at a maximal tolerable level.
  To increase the subject compliance, two measures will be implemented: timely alerts by the app (and phone calls, if needed) for performing the TEA sessions, and recording full history of therapy sessions on the device for monitoring the compliance.

SUMMARY:
This project is being completed to test the usability and safety of the Watch-Transcutaneous Electrical Acustimulation (TEA) Device.

This is a pilot study that will lead to future projects for cancer patients that may experience chemotherapy-induced symptoms.

DETAILED DESCRIPTION:
This project will include three different aims (aim three is a clinical trial) and will be funded by the National Institute of Health (NIH). In aims 1 and 2 the device hardware and device application will be developed and will not be included in this registration as these are not clinical trials. However, aim three is being registered early in the project in order to obtain the Notice of Award (NOA) funding from the NIH. Once the NOA has been obtained the registration will be updated.

ELIGIBILITY:
Inclusion Criteria:

* Participants that are willing and able to come to the clinic for two scheduled visits
* Participants are capable of understanding clinical study procedures
* Participants agree to complete the questionnaires

Exclusion Criteria:

* Participants with implanted medical devices for electrical stimulation (e.g. cardiac pacemaker)
* Those enrolled in a concurrent clinical study
* Those unable to comply with the study protocol due to a disease, psychiatric illness, alcoholism, substance abuse, geographic distance, or other factors that would place the study participant at increased risk or preclude the study participant's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Usability of the device for both groups day 3 | Day 3
  Questionnaires are administered online and there are 17 usability questions in the questionnaire. All answers use 0-to-5 scale (0 - no,1 - minor, 2 - some, 3 - considerable, 4 - major, 5 - critical) with a range of 0-85 with a higher score meaning more usable.
Number of adverse events related to the device noted on the safety questionnaire | 1-2 weeks (after baseline visit 1)
  A safety questionnaire with 3 questions about skin irritation, pain, or infection. Visit 2 is at 1-2 weeks after visit 1.
Number of Transcutaneous Electrical Acustimulation (TEA)-related adverse events for both groups 3 days | Day 3
  These will include skin irritation, pain, or infection under the Watch-TEA and tethered TEA devices after wearing each device for 3 consecutive days.
  Adverse events will be noted by the following:
  1. - Mild averse event (AE) - No treatment needed
  2. - Moderate AE - Resolved with treatment
  3. - Severe AE - Inability to carry on normal activities, required professional medical attention
  4. - Life-threatening or disabling AE
  5. - Fatal AE
Number of TEA-related adverse events for both groups 60 minutes at maximal tolerable level | Daily for 3 days
  The subjects will self-apply the TEA for 60 minutes once daily with the current amplitude set at a maximal tolerable level. Events collected will include skin irritation, pain, or infection.
  Adverse events will be noted by the following:
  1. - Mild AE - No treatment needed
  2. - Moderate AE - Resolved with treatment
  3. - Severe AE - Inability to carry on normal activities, required professional medical attention
  4. - Life-threatening or disabling AE
  5. - Fatal AE
Number of non-treatment TEA adverse events for both groups | up to 1-2 weeks (after baseline visit 1)
  Adverse events will be noted by the following:
  1. - Mild AE - No treatment needed
  2. - Moderate AE - Resolved with treatment
  3. - Severe AE - Inability to carry on normal activities, required professional medical attention
  4. - Life-threatening or disabling AE
  5. - Fatal AE

CONTACTS AND LOCATIONS:
Overall Officials: Jiande Chen, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team plans to share that information within 3 months of completing the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months of completing the study